CLINICAL TRIAL: NCT05782075
Title: Biological Monitoring by a Nurse of Post-hospital Heart Failure Patients.
Brief Title: Biological Monitoring by a Nurse for Heart Failure Patients.
Acronym: IC-SPEC
Status: Active, not recruiting | Type: Observational
Sponsor: Hôpital NOVO (Other)
Responsible Party: Sponsor
Other Study IDs: CHRD0323
Record Dates: First submitted 2023-02-22; First posted 2023-03-23 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-04

CONDITIONS: Heart Failure
Keywords: Heart failure; Biological monitoring; Heart failure nurse; Post-hospitalization
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Remote biological monitoring by a heart failure nurse — Review of biological results by a nurse (IDE) trained in heart failure monitoring, alongside the cardiologist, at S1, S2, M1, M2 and M3.

SUMMARY:
The aim of this study is to evaluate the feasibility and safety of delegating remote biological monitoring in post-hospitalization for cardiac decompensation by a heart failure nurse.

DETAILED DESCRIPTION:
Chronic heart failure is a major public health issue in France. It is the leading cause of hospitalisation in people over 65 years of age and results in many costly and potentially avoidable hospital stays. One third of patients are readmitted to hospital within 3 months of discharge.

A remote monitoring programme and natriuretic peptide monitoring during this vulnerable period can help improve patient management, reducing rehospitalisation rates, emergency room visits and mortality.

Given the increasing pressure on already limited healthcare resources, it is important to examine the delegation of care to specialist nurses, as well as their safety.

This study aims to evaluate the feasibility and safety of delegating remote biological monitoring in post-hospitalization for cardiac decompensation by a heart failure nurse.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥18 years old,
* Patient hospitalised for heart failure and discharged,
* Glomerular filtration rate at discharge > 20ml/min/1.73m²,
* Patient informed and agree to participate,
* Patient able to carry out the follow-up proposed by the cardiology department.

Exclusion Criteria:

* Cognitive disorders with Codex test category C and D,
* Barrier of the language,
* Psychiatric disorder that may interfere with treatment,
* Major surgery scheduled within 3 months,
* Excessive alcohol or drug use with no desire to withdraw
* Cardiac amyloidosis,
* Terminal heart failure,
* Patient discharged to specialised Care and Rehabilitation department,
* Any disease other than cardiac with a life expectancy of less than 1 year according to the investigator,
* Patient under guardianship,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients discharged from the cardiology department of NOVO Hospital with a heart failure episode
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-02-23 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Assessment of the concordance, appropriateness and safety of nursing decisions in post-hospitalization heart failure | At the end of the patient's follow-up, an average of 3 month
  The relevance and safety of IDE decisions will be determined by the concordance rate between the decisions made by the cardiologist and the IDE following the biological results at each check-up and after blind review by a second cardiologist

SECONDARY OUTCOMES:
Assessment of the risk of rehospitalisation in the study population between discharge and M3 | At the end of the patient's follow-up, an average of 3 month
  The risk of rehospitalization and death will be assessed, to see if a significant difference is observed between IDE decisions and cardiologist decisions, with items listed below :
  * Number of interventions initiated,
  * Number of rehospitalisation for all causes and for heart failure.
  * Number of emergency room visits for heart failure and all causes.
Assessment of the risk of death in the study population between discharge and M3 | At the end of the patient's follow-up, an average of 3 month
  The risk of death will be assessed by the rate of death for all-cause and cardiac to see if a significant difference is observed between IDE decisions and cardiologist decisions.
Impact of the organisation on patient outcomes at M3 (Brain natriuretic peptide) | At the end of the patient's follow-up, an average of 3 month
  The impact of the organisation, favourable or unfavourable, on patient outcomes will be assessed by the evolution of the following item :
  - Brain natriuretic peptide levels between discharge and three months,
Impact of the organisation on patient outcomes at M3 (New York Heart Association (NYHA)) | At the end of the patient's follow-up, an average of 3 month
  The impact of the organisation, favourable or unfavourable, on patient outcomes will be assessed by the evolution of the following item :
  - New York Heart Association (NYHA) score from discharge to three months.
Assessment of the feasibility of the patient monitoring system | At the end of the patient's follow-up, an average of 3 month
  The feasibility of the patient monitoring system will be assessed in relation to the number of biological tests not performed.
  If the number of biological tests not performed is too high, the patient monitoring system will not be validated.

CONTACTS AND LOCATIONS:
Overall Officials: Morgane Gessat, Principal Investigator — Hospital NOVO - Pontoise site
Locations (1):
- Cardiology department - Hospital NOVO - Pontoise site, Pontoise, France

REFERENCES:
- [Background] Logeart D, Isnard R, Resche-Rigon M, Seronde MF, de Groote P, Jondeau G, Galinier M, Mulak G, Donal E, Delahaye F, Juilliere Y, Damy T, Jourdain P, Bauer F, Eicher JC, Neuder Y, Trochu JN; Heart Failure of the French Society of Cardiology. Current aspects of the spectrum of acute heart failure syndromes in a real-life setting: the OFICA study. Eur J Heart Fail. 2013 Apr;15(4):465-76. doi: 10.1093/eurjhf/hfs189. Epub 2012 Nov 27. PMID 23186936
- [Background] Khan MS, Sreenivasan J, Lateef N, Abougergi MS, Greene SJ, Ahmad T, Anker SD, Fonarow GC, Butler J. Trends in 30- and 90-Day Readmission Rates for Heart Failure. Circ Heart Fail. 2021 Apr;14(4):e008335. doi: 10.1161/CIRCHEARTFAILURE.121.008335. Epub 2021 Apr 19. PMID 33866827
- [Background] Health Quality Ontario. Effect of Early Follow-Up After Hospital Discharge on Outcomes in Patients With Heart Failure or Chronic Obstructive Pulmonary Disease: A Systematic Review. Ont Health Technol Assess Ser. 2017 May 25;17(8):1-37. eCollection 2017. PMID 28638496
- [Background] Koehler F, Winkler S, Schieber M, Sechtem U, Stangl K, Bohm M, Boll H, Kim SS, Koehler K, Lucke S, Honold M, Heinze P, Schweizer T, Braecklein M, Kirwan BA, Gelbrich G, Anker SD; TIM-HF Investigators. Telemedical Interventional Monitoring in Heart Failure (TIM-HF), a randomized, controlled intervention trial investigating the impact of telemedicine on mortality in ambulatory patients with heart failure: study design. Eur J Heart Fail. 2010 Dec;12(12):1354-62. doi: 10.1093/eurjhf/hfq199. PMID 21098580
- [Background] Jourdain P, Jondeau G, Funck F, Gueffet P, Le Helloco A, Donal E, Aupetit JF, Aumont MC, Galinier M, Eicher JC, Cohen-Solal A, Juilliere Y. Plasma brain natriuretic peptide-guided therapy to improve outcome in heart failure: the STARS-BNP Multicenter Study. J Am Coll Cardiol. 2007 Apr 24;49(16):1733-9. doi: 10.1016/j.jacc.2006.10.081. Epub 2007 Apr 2. PMID 17448376